CLINICAL TRIAL: NCT06922214
Title: VT-ART-P: Ventricular Tachycardia Ablation and RadioTherapy, a Prospective Study
Brief Title: VT ART Consortium: Radioablation for Ventricular Tachycardia
Acronym: VT-ART-P
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, CELLINI FRANCESCO, Medical Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0001221/24
Record Dates: First submitted 2025-03-26; First posted 2025-04-10 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-03

CONDITIONS: Ventricular Tachycardia (VT)
Keywords: Radioablation; Ventricular Tachycardia; STAR
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Refractory ventricular tachycardia patients (Experimental): Patients with refractory VT as defined above
  1. age > 18 years
  2. ICD patients for follow-up
  3. Not eligible for heart transplantation.
  4. Prognosis not less than 1 year.
  They will have an initial assessment to verify that condition met the inclusion criteria required for participation, such as.It will be performed
  * 12-lead ECG
  * Echocardiography
  * CT scan of the chest
  * Laboratory analysis: NT proBNP, HS Troponin I
  * PMK device evaluation and clinical ECG storage.
  They will undergo stereotactic treatment on the arrhythmogenic cardiac site
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT ( 25 Gy single fractions at isodose 80%) on the area responsible of ventricular tachicardia
  Other Names: Ventricular Radioablation

SUMMARY:
The overall objective of the study is to evaluate the efficacy and safety of stereotactic radiation therapy in the non invasive ablation of ventricular tachycardia refractory to any other type treatment.

DETAILED DESCRIPTION:
By agreeing to participate in this study, the patient will undergo an initial evaluation to verify that his or her condition meets the inclusion criteria required for participation. At that visit,

* 12-lead ECG will be performed
* Echocardiography
* CT scan of the chest
* Laboratory tests: NT proBNP, HS Troponin I
* PMK device evaluation The study will have a duration of 60 months and will involve 52 patients with the same disease from which one is affected. Specifically, the total expected duration of individual subject participation in the study will be 60 months.

Participation in the study does not involve any expense for the patient or any compensation.

Participation in the study may involve some risks such as :: pericarditis, actinic pneumonia, worsening heart failure, exitus.

The following benefits can be expected from participation in this study: reduction of VT episodes compared to the pre-treatment period, reduction/total discontinuation of antiarrhythmic drugs compared to baseline (before radioablation), improvement of cardiac parameters compared to baseline : LVEF, left ventricular end-diastolic volume/diameter, end-systolic volume/diameter, RVEF and TAPSE for right ventricular function, improvement of patient's quality of life (SF-36) compared to baseline. No direct benefits may also emerge from the study, but still significant for research.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with refractory VT
2. age > 18 years
3. Patients with ICDs for follow-up
4. Ineligible for heart transplantation.
5. Prognosis of not less than 1 year
6. Ability to express autonomous consent to therapies or (in case of inability due to clinical condition) deferred consent (first indicated by the referring clinician, later expressed by the patient once recovered to autonomous condition

Exclusion Criteria:

1. Evaluation of ICD demonstrating polymorphic VT;
2. Patients with INTERMACS class greater than 4;
3. Patients with LVAD;
4. Patients with active neoplastic disease undergoing oncological treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of VT episodes | Starting from the week after treatment until 6 months later
  The primary endpoint will be The reduction in VT episodes compared with the pre-treatment period as reported by ICD assessment at follow-up within 12 months after enrollment. The number of VT episodes during the last 3 months before treatment will be compared with the number of VT episodes recorded in a 3-month period after the 'blanking period' thus during the 4th, 5th and 6th months.

SECONDARY OUTCOMES:
Change in patient management | Starting from the week after treatment until 6 months later
  Reduction in VT episodes compared with the pre-treatment period as reported by ICD query in the shortest observational period. In more detail: the number of VT episodes in the last month before treatment will be compared with the number of VT episodes recorded in the third (3rd) month after treatment.
Change in the dosage of antiarrhythmic drugs | Starting from the week after treatment until 6 months later
  Total reduction/suspension of antiarrhythmic drugs compared with baseline (before radiotherapy).
Change in cardiac parameters | Starting from the week after treatment until 6 months later
  Improvement in cardiac parameters compared with baseline: LVEF, left ventricular diastolic volume

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cellini, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Policlinico Universitario Agostino Gemelli IRCSS, Rome, RM, Italy